CLINICAL TRIAL: NCT04315818
Title: The Relation Between Macrophage Migration Inhibitory Factor (MIF) and 25(OH) Vitamin D3 Serum Levels in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Maher Abdelaziz, principal investegator, Assiut University
Other Study IDs: MIF
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: expermintal
- control group: placebo

SUMMARY:
Rheumatoid Arthritis is a chronic debilitating inflammatory autoimmune disease of unknown etiology .

DETAILED DESCRIPTION:
Although the pathogenesis of Rheumatoid Arthritis is multifactorial, the contribution of cytokines is undoubtedly pivotal in the progression of the inflammatory process. One cytokine gaining recognition for its importance in the inflammatory process is Macrophage migration inhibitory factor .

Macrophage Migration Inhibitory Factor is a multipotent cytokine involved in a broad range of functions including induction of proinflammatory mediators as well as demonstrated roles in both innate and adaptive immunity. It was originally identified in the culture medium of activated T lymphocytes as a soluble factor that inhibit random migration of macrophages .

Macrophage Migration Inhibitory Factor induces synoviocytes expression of key proinflammatory genes including TNF, IL-1, IL-6, IL-8. Moreover, it also regulates the function of endothelial cells and B cells and is implicated in the control of synoviocytes proliferation and apoptosis via direct effects on the expression of the tumor suppressor protein P53. In Rheumatoid Arthritis, increased Macrophage Migration Inhibitory Factor levels have been demonstrated in serum, synovial fluid and tissue correlating with disease activity.

Hydroxyapatite 25 vitamin D3 is a hormone primarily synthesized in human skin under the stimulation of ultraviolet radiation. Beyond its endocrine role in bone metabolism, Vitamin D3 is endowed with remarkable immunomodulatory properties. The effects of Vitamin D3 on the immune system include the enhancement of microbicidal ability of monocytes macrophages and the down-modulation of inflammatory cytokines produced by T lymphocytes.

Some epidemiological studies have reported an inverse association between serum 25(OH)vitamin D3 concentrations and Rheumatoid Arthritis disease activity and severity. In addition, some studies have reported inverse correlations between serum 25(OH)vitamin D3 and circulating inflammatory markers and cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 18 or older
* satisfying 2010 ACR/ EULAR Rheumatoid Arthritis classification criteria will be included .

Exclusion Criteria:

* Any patient with arthritis other than Rheumatoid Arthritis
* Individuals with other autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient aged 18 or older and satisfying 2010 ACR/ EULAR Rheumatoid Arthritis classification criteria will be included
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The Relation Between Macrophage Migration Inhibitory Factor (MIF) and 25(OH) Vitamin D3 Serum Levels in Rheumatoid Arthritis | october,2022
  * evaluate the role of Macrophage Migration Inhibitory Factor serum levels in Rheumatoid Arthritis and its relation with disease activity.
  * evaluate the role of 25(OH)vitamin D3 serum levels in Rheumatoid Arthritis patients and its relation to disease severity.
  * detect the relationship between Macrophage Migration Inhibitory Factor and 25(OH)vitamin D3 serum levels in Rheumatoid Arthritis patients

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Kamal, Doctor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Santos LL, Morand EF. The role of macrophage migration inhibitory factor in the inflammatory immune response and rheumatoid arthritis. Wien Med Wochenschr. 2006 Jan;156(1-2):11-8. doi: 10.1007/s10354-005-0243-8. PMID 16465610
- [Background] Kim KW, Kim HR. Macrophage migration inhibitory factor: a potential therapeutic target for rheumatoid arthritis. Korean J Intern Med. 2016 Jul;31(4):634-42. doi: 10.3904/kjim.2016.098. Epub 2016 May 12. PMID 27169879
- [Background] Llamas-Covarrubias MA, Valle Y, Navarro-Hernandez RE, Guzman-Guzman IP, Ramirez-Duenas MG, Rangel-Villalobos H, Estrada-Chavez C, Munoz-Valle JF. Serum levels of macrophage migration inhibitory factor are associated with rheumatoid arthritis course. Rheumatol Int. 2012 Aug;32(8):2307-11. doi: 10.1007/s00296-011-1951-6. Epub 2011 May 24. PMID 21607559
- [Background] Ishikawa LLW, Colavite PM, Fraga-Silva TFC, Mimura LAN, Franca TGD, Zorzella-Pezavento SFG, Chiuso-Minicucci F, Marcolino LD, Penitenti M, Ikoma MRV, Sartori A. Vitamin D Deficiency and Rheumatoid Arthritis. Clin Rev Allergy Immunol. 2017 Jun;52(3):373-388. doi: 10.1007/s12016-016-8577-0. PMID 27484684
- [Background] Bilsborrow JB, Doherty E, Tilstam PV, Bucala R. Macrophage migration inhibitory factor (MIF) as a therapeutic target for rheumatoid arthritis and systemic lupus erythematosus. Expert Opin Ther Targets. 2019 Sep;23(9):733-744. doi: 10.1080/14728222.2019.1656718. Epub 2019 Aug 20. PMID 31414920